CLINICAL TRIAL: NCT03118648
Title: Relations Between the Level Upper Limb Paresis Recovery in Output of the Hospital Unit Continued Care and Rehabilitation and Its Level of Use in Lifestyle at Three and Six Months
Brief Title: Recovery of Upper Limb Paresis at Discharge After Stroke and Its Level of Use in Activities of Daily Living 3 to 6 Months Later (Post AVC-AVQ)
Acronym: Post AVC-AVQ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2015/24
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Stroke Rehabilitation
Keywords: upper limb; functional recovery; activities of daily living

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke: * Patients over 18 years old leaving the correctional institution with orientation back home
  * First stroke deficit with non-regressive clinical expression in 24 hours
  * Independent in activities of daily living and living at home before stroke. This earlier independence is confirmed by the absence of professional carers in personal care activities
  * Proper oral understanding as measured by score 7 in the Language Screening Test (LAST) (Flamand-Roze et al, 2011)
  * No psychiatric history that led to hospitalization for more than six months
  * Written informed consent after reading the briefing note
  * Patient affiliated or beneficiary of a social security scheme.
  Interventions: Diagnostic Test: Scale Action Research Arm Test (ARAT)

INTERVENTIONS:
Diagnostic Test: Scale Action Research Arm Test (ARAT) — Measuring the functional recovery of the paretic upper limb rehabilitation outing with the scale ARAT

SUMMARY:
The aim is to reduct spontaneous use an activities of daily living of the paretic upper limb after stroke i six months after patient discharge from rehabilitation center. The level of functional recovery at rehabilitation discharge could better guide rehabilitation strategies to enhance independence and participation in daily life.

This study aims to determine, in patients after stroke, the optimal affected upper limb recovery threshold at rehabilitation discharge to predict spontaneous level of use of affected upper limb in activities of daily living, six month later.

This study is a multicentric prognostic prospective cohort study. The main prognostic variable will be the Action Arm Test (ARAT, Lyle, 1981) score at rehabilitation discharge and the predicted variable will be the Motor Activity Log - 28 (Taub et al. 1993) score at 6 months post discharge.

DETAILED DESCRIPTION:
Adults after stroke will be recruited at post-acute rehabilitation discharge. Three evaluation times will be undertaken: at discharge, three and six months after discharge. Evaluation battery will focus on the three level of the Functioning International Classification: affected upper limb level of strength, proprioception and level of functional recovery, hemineglect, depression, cognition status, and activity level by doing a standardised instrumental task of daily living, and level of participation questionnaire. General characteristics will be taken into account: Age, social status, laterality.

At six months, the spontaneous level of affected upper arm use in daily living will also be assessed using accelerometers.

As the main aim of the study is to build a prediction model, the study size is calculated to observe a minimal number of events by potentially predictive variable. We consider here 7.5 events by independent variable (Vittinghof and McCulloch, 2007) and eight independent variables. According to literature review, we estimated that 35% of adults included in this study would spontaneously use their affected upper arm in activities of daily living six months after discharge. According to these data and considering 10% of protocol deviations, we calculated that 192 subjects will have to be included in the study. The inclusion duration will be 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old leaving the correctional institution with orientation back home
* First stroke deficit with non-regressive clinical expression in 24 hours
* Independent in activities of daily living and living at home and daily activities independence before the stroke. This earlier independence is confirmed by the absence of professional carers in personal care activities (yes / no)
* Proper oral understanding as measured by score 7 in the language screening test LAST (Flamand-Roze et al, 2011)
* No psychiatric history that led to hospitalization for more than six months
* Patient has given its consent within the period provided after reading the briefing note
* Patient affiliated or beneficiary of a social security scheme.

Exclusion Criteria:

* Lack of minimum functional motor recovery in paretic upper limb allowing the patient to go put hand to his mouth and to realize do a 45 degrees abduction with the paretic upper limb.
* Barthel Index score (BI) less than or equal to 40. It is suggested in the literature that a score less than or equal to 40 is a key score of total dependence
* Persistent severe hemineglect (bells test score > 6).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible to participate in the study will be adults who have experienced a first stroke and are about to leave the rehabilitation facility for their home. These people should have a good oral comprehension. They must not have a psychiatric history with hospitalization of more than 6 months. They must have been independent in the activities of daily life before their stroke. They must be affiliated to a social security scheme, be willing to participate in the study and not participate in another research.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Motor Activity | Month 6
  Score of Motor Activity Log scale

SECONDARY OUTCOMES:
Action Arm | Day 0
  Score of Action Research Arm Test scale
Action Arm | Day 180
  Score of Action Research Arm Test scale
Cognitive abilities | Day 0
  Score with kettle test
Cognitive abilities | Day 180
  Score with kettle test
"Mesure des HAbitudes de VIE" (MHAVIE) | Day 0
  Score of "Mesure des HAbitudes de VIE" scale (MHAVIE)
"Mesure des HAbitudes de VIE" (MHAVIE) | Day 180
  Score of "Mesure des HAbitudes de VIE" scale (MHAVIE)
"Montreal Cognitive Assessment" (MoCA) | Day 0
  Score of "Montreal Cognitive Assessment" (MoCA)
"Montreal Cognitive Assessment" (MoCA) | Day 180
  Score of "Montreal Cognitive Assessment" (MoCA)
Aphasic Depression Rating (ADRS) | Day 0
  Score of Aphasic Depression Rating Scale (ADRS)
Aphasic Depression Rating (ADRS) | Day 180
  Score of Aphasic Depression Rating Scale (ADRS)
Unilateral spatial neglect (NSU) in the vicinity of extrapersonal space | Day 0
  Score of "Bell test (test de barrage des cloches)"
Unilateral spatial neglect (NSU) in the vicinity of extrapersonal space | Day 180
  Score of "Bell test (test de barrage des cloches)"

CONTACTS AND LOCATIONS:
Overall Officials: Eric SORITA, PhD, Principal Investigator — University Hospital, Bordeaux; Paul PEREZ, MD, Study Chair — Unité de Soutien Méthodologique à la Recherche Clinique et Epidémiologique du CHU de Bordeaux
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lyle RC. A performance test for assessment of upper limb function in physical rehabilitation treatment and research. Int J Rehabil Res. 1981;4(4):483-92. doi: 10.1097/00004356-198112000-00001. No abstract available. PMID 7333761
- [Background] Taub E, Miller NE, Novack TA, Cook EW 3rd, Fleming WC, Nepomuceno CS, Connell JS, Crago JE. Technique to improve chronic motor deficit after stroke. Arch Phys Med Rehabil. 1993 Apr;74(4):347-54. PMID 8466415
- [Background] Vittinghoff E, McCulloch CE. Relaxing the rule of ten events per variable in logistic and Cox regression. Am J Epidemiol. 2007 Mar 15;165(6):710-8. doi: 10.1093/aje/kwk052. Epub 2006 Dec 20. PMID 17182981
- [Background] Uswatte G, Giuliani C, Winstein C, Zeringue A, Hobbs L, Wolf SL. Validity of accelerometry for monitoring real-world arm activity in patients with subacute stroke: evidence from the extremity constraint-induced therapy evaluation trial. Arch Phys Med Rehabil. 2006 Oct;87(10):1340-5. doi: 10.1016/j.apmr.2006.06.006. PMID 17023243
- [Background] Veerbeek JM, Kwakkel G, van Wegen EE, Ket JC, Heymans MW. Early prediction of outcome of activities of daily living after stroke: a systematic review. Stroke. 2011 May;42(5):1482-8. doi: 10.1161/STROKEAHA.110.604090. Epub 2011 Apr 7. PMID 21474812
- [Background] Rand D, Eng JJ. Predicting daily use of the affected upper extremity 1 year after stroke. J Stroke Cerebrovasc Dis. 2015 Feb;24(2):274-83. doi: 10.1016/j.jstrokecerebrovasdis.2014.07.039. Epub 2014 Dec 18. PMID 25533758